CLINICAL TRIAL: NCT01017354
Title: Monthly Vitamin D to Improve Vitamin D Status and Maintain Function in Pre-frail Older Individuals Living at Home
Brief Title: Zurich Disability Prevention Trial
Acronym: ZDPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KEK39/09; 2009DR2248 (Other: Swissmedic (Swiss Agency for Therapeutic Products))
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Community-dwelling Seniors; History of a Fall in the Previous 12 Months
Keywords: vitamin D; function; falls; 25-hydroxyvitamin D; disability
MeSH Terms: interventions — Calcifediol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High-dose vitamin D3 (Experimental): monthly high-dose vitamin D3 supplement dose (60'000 IU/month, equivalent to 2000 IU daily)
  Interventions: Dietary Supplement: ViDe3 (CH)
- standard vitamin D + 25(OH)D (Experimental): standard vitamin D3 supplement dose combined with 25(OH)D (24'000 IU/month, equivalent to 800 IU daily PLUS 300 mcg 25(OH)D, equivalent to 10 mcg per day)
  Interventions: Drug: Hidroferol® (ES)
- standard vitamin D (Active Comparator): standard vitamin D3 supplement dose (24'000 IU/month, equivalent to 800 IU daily)
  Interventions: Dietary Supplement: ViDe3 (CH)

INTERVENTIONS:
Drug: Hidroferol® (ES) — 24000 IU vitamin D3 orally and once per month plus 300 mcg 25(OH)D orally and once per month
  Arms: standard vitamin D + 25(OH)D
Dietary Supplement: ViDe3 (CH) — 60000 vitamin D3 orally and once per month
  Arms: High-dose vitamin D3
Dietary Supplement: ViDe3 (CH) — 24000 Vitamin D3 orally and once per month
  Arms: standard vitamin D

SUMMARY:
This project was designed to optimizing vitamin D status in prefrail seniors age 70+ living at home and prevent their functional decline. We test 3 arms of monthly vitamin D supplementation. Intermittent dosing will improve adherence and simplify vitamin D supplementation.

DETAILED DESCRIPTION:
We propose a double-blind, randomized controlled trial to test the effectiveness of a

1. Active I (n=70): monthly high-dose vitamin D3 supplement dose (60'000 IU/month, equivalent to 2000 IU daily),
2. Active II (n=70): or a monthly standard vitamin D3 supplement dose combined with 25(OH)D (24'000 IU/month, equivalent to 800 IU daily PLUS 300 mcg 25(OH)D, equivalent to 10 mcg per day)
3. Control (n=70): compared to a standard vitamin D3 supplement dose (24'000 IU/month, equivalent to 800 IU daily)

All individuals will be advised to consume calcium from natural food sources in a daily dose of 600-800 mgs a day, including milk products. Maximal intake of supplemental calcium is restricted to 250 mg per day.

ELIGIBILITY:
Inclusion criteria:

* Age 70+
* Fall in the last 12 months before screening (with or without a fracture)
* Living at home (community-dwelling)
* Men or women
* Mobile with or without walking aid - have to be able to use public transportation to attend the clinical visits at the trial centre
* Score of at least 27 at the screening Folstein Mini Mental test + normal clock test
* Patient understands the study procedures, alternative treatments available and risks involved with the study, and voluntarily agrees to participate by giving a written informed consents.
* Patient meets the entry minimal requirements based on routine clinical laboratory safety screening tests and the Folstein mini mental status (score 27+ required) performed at the Screening Visit.
* Patient is willing to perform all study tests, attend all required office visits, and provide blood and urine samples.

Exclusion criteria:

* Serum calcium adjusted for albumin of > 2.6 nmol/l
* Pathologic fracture in the last year (except for fractures due to osteoporosis)
* Chemo therapy / Radiation due to cancer in the last year
* Treatment which has an effect on bone metabolism (e.g. bisphosphonate, PTH, calcitonin, chronic cortisone intake > XYmg/day for more than XY month/years (except for inhalation and sporadic infiltration))
* Oral vitamin D intake of more than 800 IU per day
* Unwilling to stop calcium supplementation and vitamin D supplementation during the trial (maximal calcium supplement intake 250mg/d; no additional vitamin D supplementation)
* Severe visual or hearing impairment
* Unwilling or unable to take study medication
* Diseases with a risk of recurrent falling (e.g. Parkinson's disease/syndrome, Hemiplegia after stroke, symptomatic stenosis of the spinal canal, polyneuropathy, epilepsy, recurring vertigo, recurring syncope)
* BMI >= 40
* Estimated creatinine clearance < 15 ml/min (estimated Creatinine Clearance Cockcroft and Gault)
* Malabsorption syndrome (celiac diseases, inflammatory bowl disease)
* Diseases that may enhance serum calcium: sarcoidosis, lymphoma, primary hyperparathyroidism
* kidney stone in the last 10 years
* Abnormal indices of calcium metabolism, uncontrolled hypocalcemia.
* Patient heavily consumes alcohol containing products defined as greater than (>) 3 drinks (beer, wine, or distilled spirits) of alcoholic beverages per day.
* Patient is unlikely to adhere to the study procedures, to keep appointments, or is planning to relocate during the study.
* Patients who are planning a stay in a "sunny" location (e.g. winter sun resort) for more than two months per year
* Medication which has an effect on 25-hydroxyvitamin D level (e.g. certain anticonvulsants (e.g. Phenobarbital, Carbamazepin, Phenytoin))
* M. Paget (Ostitis deformans)
* inflammatory arthritis (e.g. rheumatoid arthritis, reiter syndrome, psoriasis arthritis)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
functional decline (proportion of individuals with functional decline based on binary repeated measure assessment across 4 lower extremity tests) | 6 and 12 months
Improving 25-hydroxyvitamin D levels in late winter and late summer - Percent of individuals reaching desirable 25-hydroxyvitamin D levels of at least 75 nmol/l in late winter and in late summer | 6 and 12 months

SECONDARY OUTCOMES:
Safety at baseline, 2 weeks, 6 months, 12 months • Serum calcium adjusted for albumin • Serum creatinine • Urinary calcium/creatinine ratio | 2 weeks, 6 months, 12 months
Balance/Gait while walking combined with a cognitive task | 12 months
Short Physical Performance Test Battery | 6 months, 12 months
Timed 4 m walk | 6 months, 12 months
Musculoskeletal pain assessed with the McGill pain map | 6 months and 12 months
systolic and diastolic blood pressure, heart rate | 6 month and 12 months
Rate of falls, all, injurious falls (diary, monthly phone calls, and hotline) | 12 months
grip strength | 6 months and 12 months
Bone density at the spine and hip, whole body | 6 months and 12 months
incident vertebral fractures (iDXA morphometry) | 12 months
muscle mass, incident sarcopenia | 6 and 12 months
Health care utilization: in collaboration with insurance companies for outpatient and inpatient health care costs. | 12 months
Quality of life (SF 12 / EuroQuol) | 6 months and 12 months
Rate of hospital admission (fall-related injury, infections, other) | 12 months
Serum N-telopeptides and other markers of bone remodeling | 6 months and 12 months
Upper and lower respiratory tract infections, any infections, infections that lead to inpatient care | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff Ferrari, MD, MPH, Principal Investigator — University Hospital Zurich, Centre on Aging and Mobility
Locations (1):
- University Hospital Zurich, Centre on Aging and Mobility, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Braendle K, Egli A, Bischoff-Ferrari H, Freystaetter G. Does living alone influence fall risk among Swiss older adults aged 60+? A pooled observational analysis of three RCTs on fall prevention. BMJ Open. 2024 May 20;14(5):e081413. doi: 10.1136/bmjopen-2023-081413. PMID 38772577
- [Derived] Bischoff-Ferrari HA, Dawson-Hughes B, Orav EJ, Staehelin HB, Meyer OW, Theiler R, Dick W, Willett WC, Egli A. Monthly High-Dose Vitamin D Treatment for the Prevention of Functional Decline: A Randomized Clinical Trial. JAMA Intern Med. 2016 Feb;176(2):175-83. doi: 10.1001/jamainternmed.2015.7148. PMID 26747333